CLINICAL TRIAL: NCT00968669
Title: A Phase 2b, Randomized Study to Evaluate the Efficacy and Safety of Subcutaneous MEDI-528 in Adults With Uncontrolled Asthma
Brief Title: A Study to Evaluate the Effectiveness and Safety of MEDI-528 in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP198
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Results first posted 2014-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — enokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MEDI528 30 mg (Experimental): MEDI-528 at a dose of 30 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Interventions: Biological: MEDI528 30 mg
- MEDI528 100 mg (Experimental): MEDI-528 at a dose of 100 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Interventions: Biological: MEDI528 100 mg
- MEDI528 300 mg (Experimental): MEDI-528 at a dose of 300 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Interventions: Biological: MEDI528 300 mg
- Placebo (Experimental): Placebo administered as a subcutaneous injection every 2 weeks for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: MEDI528 30 mg — MEDI-528 at a dose of 30 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Arms: MEDI528 30 mg
Biological: MEDI528 100 mg — MEDI-528 at a dose of 100 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Arms: MEDI528 100 mg
Biological: MEDI528 300 mg — MEDI-528 at a dose of 300 mg administered as a subcutaneous injection every 2 weeks for 24 weeks
  Arms: MEDI528 300 mg
Other: Placebo — Placebo administered as a subcutaneous injection every 2 weeks for 24 weeks
  Arms: Placebo

SUMMARY:
To study the effectiveness and safety of multiple-doses of MEDI-528 on asthma control in adult participants with uncontrolled, moderate-to-severe, persistent asthma.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the effect of multiple-dose subcutaneous (SC) administration of MEDI-528 on asthma control in adults with uncontrolled, moderate-to-severe, persistent asthma.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria:

1. Male or female
2. Age 18 through 65 years at the time of screening
3. Written informed consent and any locally required authorization obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
4. Female subjects of childbearing potential who are sexually active with non-sterilized male partner must use adequate contraception from screening through the end of the study. An acceptable method of contraception is defined as one that has no higher than a 1% failure rate. Sustained abstinence is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception

   1. Non-sterilized males who are sexually active with a female of child-bearing potential must use adequate contraception from screening through the end of the study
   2. Females or female partners not of childbearing potential must have been surgically sterilized (eg, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or postmenopausal (defined as at least 1 year since last regular menses)
   3. Sterilized males must be at least 1-year post vasectomy and have obtained documentation of the absence of sperm in the ejaculate
5. Weight ≥ 45 kg but ≤ 120 kg and body mass index (BMI) between 18 and 35 kg/m2
6. Physician-diagnosed asthma by medical chart
7. Currently taking inhaled corticosteroids (ICS) or is a candidate to receive ICS per Expert Panel Report (EPR)-3
8. Pre-bronchodilator forced expiratory volume in 1 second (FEV1) value ≥ 40% at Day -28 and Day 1
9. A post-bronchodilator increase in FEV1 and/or FVC ≥ 12% and ≥ 200 mL at Day -28 OR meeting any one of the following criteria:

   1. Proof of post-bronchodilator reversibility of airflow obstruction ≥ 12% documented within 36 months prior to randomization or proof of a positive response to a methacholine challenge documented within 36 months prior to randomization; OR
   2. Proof of partial reversibility of ≥ 8% to < 12% improvement in post-bronchodilator FEV1 on Day -28 and achievement of ≥ 12% reversibility at a second time between Day -27 and Day -15; OR
   3. If a) and b) are not met and all other inclusion/exclusion criteria are met, subjects with a FEV1 of ≥ 1.5 L and ≥ 60% on Day -14 will be eligible to undergo a methacholine challenge. If the subject achieves a positive response to this methacholine challenge, then this criterion is met
10. Uncontrolled asthma consistent with EPR-3. In the 28 days before screening, subjects should have a history of one or more of the following:

    * Daytime asthma symptoms ≥ 2 days/week
    * Nighttime awakening ≥ 1 night/week
    * Albuterol/salbutamol use ≥ 2 days/week
11. An Asthma Control Questionnaire (ACQ) score ≥ 1.5 at Day -28 and at Day 1.
12. At least one asthma exacerbation in the 12 months before screening that required intake of systemic corticosteroids after an unscheduled medical encounter or as agreed with a physician based on an asthma action plan that defines when oral steroids can be taken by the subject
13. Ability and willingness to complete the follow-up period through Day 323 as required by the protocol.

Exclusion Criteria

Any of the following would exclude the subject from participation in the study:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
2. Concurrent enrollment in another clinical study
3. Employees of the clinical study site or any other individuals involved with the conduct of the study, or immediate family members of such individuals
4. Known history of allergy or reaction to any component of the investigational product formulation
5. History of anaphylaxis to other biologic therapy
6. Lung disease other than asthma (eg, chronic obstructive pulmonary disease [COPD], cystic fibrosis)
7. Severe depression as measured by a depression score > 15 on the Hospital Anxiety and Depression Scale (HADS) at either Day-28 or Day 1.
8. History of suicidal behavior in the previous 3 years as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) at Day -28.
9. Acute illness other than asthma at the screening and randomization visits
10. History of an active infection within 28 days before and during the screening period, or evidence of clinically significant active infection, including ongoing chronic infection
11. History of ingestion of untreated water in a location known to be infected with parasites, resulting in acute or chronic diarrhea; history of recent travel to areas where parasite infestations are endemic within 6 months before screening; or a diagnosis of parasitic infection within 6 months before screening
12. Use of immunosuppressive medication (except oral prednisone up to a dose of 20 mg every other day or equivalent [eg, 10 mg a day or 5 mg twice a day] and inhaled and topical corticosteroids) within 28 days before randomization
13. Receipt of immunoglobulin or blood products within 28 days before randomization
14. Plans to donate blood during the entire study period
15. Donated blood or has had a blood transfusion within 28 days before screening
16. Receipt of any non-biological study drugs or interventional therapy (including surgical procedures) within 28 days of the first dose of investigational product in this study
17. Receipt of any biologicals including MEDI-528 within 5 half-lives before the first dose of investigational product in this study
18. History of any known immunodeficiency disorder
19. A positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history and/or subject's verbal report
20. A positive human immunodeficiency virus test or is taking antiretroviral medications, as determined by medical history and/or subject's verbal report
21. A live attenuated vaccination received within 28 days before screening
22. History of clinically significant abnormality on electrocardiogram (ECG) in the opinion of the investigator
23. Breastfeeding or lactating
24. History of treatment for alcohol or drug abuse within the past year
25. History suggestive of COPD or of tobacco smoking ≥ 10 pack-years
26. Evidence of any uncontrolled systemic disease upon physical examination
27. History of cancer, apart from basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy ≥ 1 year before Day 1 or other malignancies treated with apparent success with curative therapy ≥ 5 years before screening
28. Any noninfectious disease involving multiple organs (eg, cystic fibrosis, systemic lupus erythematosus, hemophilia, multiple sclerosis, etc.) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results
29. Individuals who are legally institutionalized

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2009-12; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Oh, M.D., Study Director — MedImmune LLC
Locations (53):
- United States (24):
  - Research Site, Pell City, Alabama
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Centennial, Colorado
  - Research Site, Colarado Springs, Colorado
  - Research Site, Thornton, Colorado
  - Research Site, Waterbury, Connecticut
  - Research Site, Kissimmee, Florida
  - Research Site, Normal, Illinois
  - Research Site, Overland Park, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Baltimore, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Minneapolis, Minnesota
  - Research Site, Omaha, Nebraska
  - Research Site, Mount Laurel, New Jersey
  - Research Site, Sylvania, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Lincoln, Rhode Island
  - Research Site, Greenville, South Carolina
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas
- Argentina (6):
  - Research Site, Buenos Aire, Buenos Aires F.D.
  - Research Site, Ciudad Autonoma Bs As, Buenos Aires F.D.
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Buenos Aires
  - Research Site, Ciudad de Buenos Aire
- Brazil (4):
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Florianópolis, Santa Catarina
  - Research Site, Santo André
  - Research Site, São Paulo
- Canada (7):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- Colombia (3):
  - Research Site, Bogota DC, Cundinamarca
  - Research Site, Bogota, Cundinamarca
  - Research Site, Bogotá D.C., Cundinamarca
- Research Site, San Francisco de Dos Ríos, Provincia de San José, Costa Rica
- Research Site, Panama City, Panama
- Peru (2):
  - Research Site, Lima, Lima Province
  - Research Site, Jesus Maria, Lima region
- Philippines (3):
  - Research Site, Lipa City, Batangas
  - Research Site, Iloilo City, Iloilo
  - Research Site, Quezon City, National Capital Region
- Taiwan (2):
  - Research Site, Kaohsiung City
  - Research Site, Taoyuan District

REFERENCES:
- [Derived] Oh CK, Leigh R, McLaurin KK, Kim K, Hultquist M, Molfino NA. A randomized, controlled trial to evaluate the effect of an anti-interleukin-9 monoclonal antibody in adults with uncontrolled asthma. Respir Res. 2013 Sep 19;14(1):93. doi: 10.1186/1465-9921-14-93. PMID 24050312
- [Derived] Lloyd CM, Hessel EM. Functions of T cells in asthma: more than just T(H)2 cells. Nat Rev Immunol. 2010 Dec;10(12):838-48. doi: 10.1038/nri2870. Epub 2010 Nov 9. PMID 21060320

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 329 participants was randomized into the study, but 2 participants (1 in the MEDI-528 30 mg arm and 1 in the MEDI-528 300 mg arm) were randomized by mistake as they were screen failures. Therefore, a total of 327 participants were correctly randomized into the study.
Period: Overall Study
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Started | 82 | 81 | 83 | 81
Completed | 64 | 63 | 72 | 72
Not Completed | 18 | 18 | 11 | 9
Not completed — Lost to Follow-up | 5 | 2 | 1 | 4
Not completed — Withdrawal by Subject | 9 | 7 | 5 | 3
Not completed — Pregnancy | 0 | 0 | 2 | 0
Not completed — AE | 1 | 0 | 0 | 0
Not completed — AE-TRANSITIONAL CELL TUMOR IN BLADDER | 0 | 0 | 0 | 1
Not completed — DID NOT MEET EXCLUSION CRITERIA | 1 | 0 | 0 | 0
Not completed — DUE TO REPEATED ASTHMA EXACERBATIONS | 1 | 0 | 0 | 0
Not completed — EARLY DISCONTINUED ON 10-DEC-2010 | 0 | 0 | 1 | 0
Not completed — EARLY WITHDRAWAL | 0 | 1 | 0 | 0
Not completed — ERROR IN HADS ADMINISTRATION | 0 | 0 | 1 | 0
Not completed — INEGIBILITY TO PERFORM VISIT | 1 | 0 | 0 | 0
Not completed — PATIENT RECEIVE ORAL PREDNISONE | 0 | 1 | 0 | 0
Not completed — PATIENT WAS ENROLLED BY MISTAKE | 0 | 1 | 0 | 0
Not completed — PATIENT WAS RANDOMIZED BY MISTAKE | 0 | 1 | 0 | 0
Not completed — PATIENT WILL BE WORKING ABROAD | 0 | 1 | 0 | 0
Not completed — SPONSOR DECISION | 0 | 1 | 0 | 0
Not completed — SUBJECT COMPLETED SAFETY FOLLOW-UP | 0 | 0 | 1 | 0
Not completed — SUBJECT DID NOT MEET ACQ REQUIREMENT | 0 | 1 | 0 | 0
Not completed — SUBJECT INCARCERATED | 0 | 1 | 0 | 0
Not completed — SUBJECT WAS RANDOMIZED IN ERROR | 0 | 1 | 0 | 0
Not completed — WITHDRAWN DUE TO PREDNISONE USE | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg | Total
Number analyzed (Participants) | 82 | 81 | 83 | 81 | 327
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.6 (11.6) | 41.8 (11.1) | 45.1 (11.6) | 41.5 (12.3) | 43.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 55 | 62 | 55 | 225
  Male | 29 | 26 | 21 | 26 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change at Day 92 From Baseline in Mean Asthma Control Questionnaire (ACQ) Scores (Intent-toTreat Analysis)
Description: Change at Day 92 from baseline (Day 1, prior to dosing) in mean ACQ scores in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Day 92
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 (n=81, 83, or 81, respectively) or placebo (n=82) groups.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Scores on a scale | -1.23 (0.95) | -1.10 (1.11) | -1.26 (1.02) | -1.31 (1.07)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.435, ANOVA; Missing mean ACQ scores at Day 92 was imputed by last observation carried forward
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.828, ANOVA; Missing mean ACQ scores at Day 92 was imputed by last observation carried forward
Statistical Analysis 3: Comparison: MEDI528 300 mg; Test type: Superiority or Other; p = 0.628, ANOVA; Missing mean ACQ scores at Day 92 was imputed by last observation carried forward

2. Secondary Outcome: Weighted Asthma Exacerbation Rate Through Day 92 (Intent-to-Treat Analysis)
Description: Weighted asthma exacerbation rate (total number of exacerbation rate in each group per total duration of participant-year follow-up in each group) between Day 1 and Day 92 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 92
Population: All participants who were randomized and received at least one dose of investigational product (30, 100, or 300 mg MEDI-528 or placebo)
Measure: Number (95% Confidence Interval); unit: Exacerbations per participant year
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Exacerbations per participant year | 0.53 (0.96) [0.27 to 0.96] | 0.82 (1.15) [0.47 to 1.33] | 0.33 [0.13 to 0.68] | 0.39 [0.17 to 0.77]
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.271, Pairwise Poisson Regression
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.319, Pairwise Poisson Regression
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.502, Pairwise Poisson Regression

3. Secondary Outcome: Weighted Asthma Exacerbation Rate Through Day 176 (Intent-to-Treat Analysis)
Description: Weighted asthma exacerbation rate (total number of exacerbation rate in each group per total duration of participant-year follow-up in each group) between Day 1 and Day 176 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 176
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Exacerbations per participant year
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Exacerbations per participant year | 0.58 (0.96) [0.36 to 0.88] | 0.64 (1.15) [0.40 to 0.96] | 0.28 [0.14 to 0.50] | 0.58 [0.36 to 0.88]
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.756, Pairwise Poisson Regression
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.047, Pairwise Poisson Regression
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 1.000, Pairwise Poisson Regression

4. Secondary Outcome: Proportion of Participants Experiencing at Least One Asthma Exacerbation Through Day 92 (Intent-to-Treat Analysis)
Description: The proportion of participants that experienced at least one asthma exacerbation between Day 1 and Day 92 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 92
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Participants | 8 (0.15) [0.36 to 0.88] | 14 (0.14) [0.36 to 0.88] | 5 | 7
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.1764, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.4031, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact

5. Secondary Outcome: Proportion of Participants Experiencing at Least One Asthma Exacerbation Through Day 176 (Intent-to-Treat Analysis)
Description: The proportion of participants that experienced at least one asthma exacerbation between Day 1 and Day 176 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 176
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Participants | 16 (0.15) [0.36 to 0.88] | 17 (0.14) [0.36 to 0.88] | 8 | 15
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.8475, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.0811, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 1.0000, Fisher Exact

6. Secondary Outcome: Time to First Asthma Exacerbation Through Day 92 (Intent-to-Treat Analysis)
Description: Time to first asthma exacerbation between Day 1 and Day 92 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 92
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Day | NA (2.10) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (3.38) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (2.14) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (2.27) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached.
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.144, Log Rank; Stratified by atopic asthma and steroid use; Hazard Ratio (HR) = 1.938
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.395, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.618
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.863, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.899

7. Secondary Outcome: Time to First Asthma Exacerbation Through Day 176 (Intent-to-Treat Analysis)
Description: Time to first asthma exacerbation between Day 1 and Day 176 in pariticpants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). An exacerbation was defined as a progressive increase of asthma symptoms AND a reduction of 20% or more in peak expiratory flow (PEF) or forced expiratory volume in 1 second (FEV1) from baseline (Day 1, prior to dosing) or best previously measured value prior to the current event that did not resolve after the initiation of rescue medications; and results in a prescription for/or administration of systemic corticosteroid burst therapy by the investigator or health care provider. An exacerbation event was considered resolved when the subject's asthma symptoms diminished and PEF or FEV1 return to greater than 80% of baseline for 7 or more days after completion of systemic corticosteroid burst therapy.
Time Frame: Days 1 - 176
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Day | NA (5.30) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (7.15) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (4.70) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached. | NA (5.40) [NA to NA] — Too few events; time to median time to first asthma exacerbation was not reached.
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.717, Log Rank; Stratified by atopic asthma and steroid use; Hazard Ratio (HR) = 1.162
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.070, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.467
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.934, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.955

8. Secondary Outcome: Change at Day 176 From Baseline in Mean Asthma Control Questionnaire Scores (Intent-to-Treat Analysis)
Description: Change at Day 176 from baseline (Day 1, prior to dosing) in mean ACQ scores in participants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Day 176
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had ACQ data available on Day 176.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Scores on a scale | -1.27 (1.17) | -1.32 (1.23) | -1.46 (1.07) | -1.45 (1.08)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.813, ANOVA
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.290, ANOVA
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.303, ANOVA

9. Secondary Outcome: Proportion of Participants Achieving Mean Asthma Control Questionnaire (ACQ) Scores at Day 92 of < or = 0.75, > 0.75 to < 1.5, and > or = 1.5 (Intent-to-Treat Analysis)
Description: Proportion of participants achieving mean ACQ scores of < or = 0.75, > 0.75 to < 1.5, and > or = 1.5 at Day 92 in participants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Day 92
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had ACQ data available on Day 92.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Participants
  < or = 0.75 | 17 | 17 | 17 | 22
  > 0.75 and < 1.5 | 23 | 21 | 22 | 16
  > or = 1.5 | 42 | 43 | 44 | 43
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg vs MEDI528 100 mg vs MEDI528 300 mg; Combined MEDI-528 treatment was compared to placebo; Test type: Superiority or Other; p = 0.764, Fisher Exact

10. Secondary Outcome: Proportion of Participants Achieving Mean Asthma Control Questionnaire (ACQ) Scores at Day 176 of < or = 0.75, > 0.75 to < 1.5, and > or = 1.5 (Intent-to-Treat Analysis)
Description: Proportion of participants achieving mean ACQ scores of < or = 0.75, > 0.75 to < 1.5, and > or = 1.5 at Day 176 in participants receiving 30, 100, or 300 mg MEDI-528 versus placebo (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Day 176
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Participants
  < or = 0.75 | 25 | 29 | 24 | 25
  > 0.75 and < 1.5 | 19 | 18 | 18 | 20
  > or = 1.5 | 38 | 34 | 41 | 36
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg vs MEDI528 100 mg vs MEDI528 300 mg; Combined MEDI-528 treatment was compared to placebo; Test type: Superiority or Other; p = 0.986, Fisher Exact

11. Secondary Outcome: Time to First Observed Mean Asthma Control Questionnaire (ACQ) Change From Baseline > or = 0.5 Through Day 92 (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the time to first observed mean ACQ change from baseline (Day 1, prior to dosing) > or = 0.5 through Day 92 (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Days 1 - 92
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had ACQ data through Day 92.
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Day | 15.0 (2.62) [15.0 to 22.0] | 17.0 (2.93) [15.0 to 21.0] | 20.0 (2.67) [15.0 to 23.0] | 20.0 (2.89) [15.0 to 27.0]
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.7171, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.955
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.6219, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.942
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.6182, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.909

12. Secondary Outcome: Time to First Observed Mean Asthma Control Questionnaire (ACQ) Change From Baseline > or = 0.5 Through Day 176 (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the time to first observed mean ACQ change from baseline (Day 1, prior to dosing) > or = 1.5 Through Day 176 (Intent-to-Treat Analysis). The 6-item ACQ is a participant-reported questionnaire assessing asthma symptoms (night-time waking, symptoms on waking, activity limitation, shortness of breath, wheezing) and daily rescue bronchodilator use. Participants were asked to recall how their asthma had been during the previous week. Questions were weighted equally and scored from 0 (totally controlled) to 6 (severely uncontrolled). The mean ACQ score is the mean of the responses. Mean scores of ≤ 0.75 indicate well-controlled asthma, scores between 0.76 and < 1.5 indicate partly controlled asthma, and a score ≥ 1.5 indicates uncontrolled asthma. Individual changes of at least 0.5 are considered to be clinically meaningful.
Time Frame: Days 1 - 176
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had ACQ data through Day 176.
Measure: Median (95% Confidence Interval); unit: Day
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Day | 15.0 (4.07) [15.0 to 22.0] | 17.0 (4.57) [15.0 to 21.0] | 20.0 (3.63) [15.0 to 23.0] | 20.0 (4.70) [15.0 to 27.0]
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.7120, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.952
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.5086, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.928
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.5184, Log Rank; Stratified by atopic asthma status and steroid use; Hazard Ratio (HR) = 0.887

13. Secondary Outcome: Change at Day 92 From Baseline in Forced Expiratory Volume in One Second (FEV1) (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the mean change at Day 92 from baseline (Day 1, prior to dosing) in FEV1.
Time Frame: Day 92
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 (n=81, 83, or 81, respectively) or placebo (n=82) groups who had FEV1 data available at Day 92 (n=62, 73, or 72 for 30, 100, or 300 mg MEDI-528, respectively, and n=67 for placebo).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 67 | 62 | 73 | 72
Liters | 0.033 (0.326) | 0.045 (0.327) | 0.048 (0.230) | 0.097 (0.290)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.837, Two-sample t-test
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.756, Two-sample t-test
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.224, Two-sample t-test

14. Secondary Outcome: Change at Day 176 From Baseline in Forced Expiratory Volume in One Second (FEV1) (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the mean change from baseline (Day 1, prior to dosing) in FEV1 at Day 176
Time Frame: Day 176
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 (n=81, 83, or 81, respectively) or placebo (n=82) groups who had FEV1 data available at Day 176 (n=67, 75, or 73 for 30, 100, or 300 mg MEDI-528, respectively, and n=69 for placebo).
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 69 | 67 | 75 | 73
Liters | 0.044 (0.367) | -0.005 (0.324) | 0.055 (0.299) | 0.047 (0.290)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg; Test type: Superiority or Other; p = 0.409, Two-sample t-test
Statistical Analysis 2: Comparison: Placebo vs MEDI528 100 mg; Test type: Superiority or Other; p = 0.847, Two-sample t-test
Statistical Analysis 3: Comparison: Placebo vs MEDI528 300 mg; Test type: Superiority or Other; p = 0.968, Two-sample t-test

15. Secondary Outcome: Proportion of Participants Who Had a Asthma Quality of Life Questionnaire - Standard (AQLQ[S]) Assessment Response at Day 85 (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the proportion of participants who had an AQLQ(S) assessment response (defined as an improvement of at least 0.5 score in AQLQ[S]) at Day 85 (Intent-to-Treat Analysis). The AQLQ(S) is a 32-item questionnaire that measures the health related quality of life experienced by asthma patients. In the study, participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean response to all questions. Individual improvement in the overall score of 0.5 has been identified as the minimally important difference, with score changes > 1.5 identified to be large meaningful differences.
Time Frame: Day 85
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had AQLQ(S) data at Day 85 (n=69, 63, 76, and 68 for placebo, 30, 100, and 300 mg MEDI-528, respectively).
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 69 | 63 | 76 | 68
Participants | 53 (57.871) | 43 (60.584) | 52 (53.110) | 49 (55.339)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg vs MEDI528 100 mg vs MEDI528 300 mg; Combined MEDI-528 dose groups versus placebo; Test type: Superiority or Other; p = 0.208, Fisher Exact

16. Secondary Outcome: Proportion of Participants Who Had a Asthma Quality of Life Questionnaire - Standard (AQLQ[S]) Assessment Response at Day 176 (Intent-to-Treat Analysis)
Description: Effect of MEDI-528 (30, 100, or 300 mg) versus placebo on the proportion of participants who had an AQLQ(S) assessment response at Day 176 (Intent-to-Treat Analysis). The AQLQ(S) is a 32-item questionnaire that measures the health related quality of life experienced by asthma patients. In the study, participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score is calculated as the mean response to all questions. Individual improvement in the overall score of 0.5 has been identified as the minimally important difference, with score changes > 1.5 identified to be large meaningful differences.
Time Frame: Day 176
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo group (n=82) who had AQLQ(S) data at Day 176 (n=62, 58, 64, and 60 for placebo, 30, 100, and 300 mg MEDI-528, respectively).
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 62 | 58 | 64 | 60
Participants | 50 (57.871) | 42 (60.584) | 48 (53.110) | 46 (55.339)
Statistical Analysis 1: Comparison: Placebo vs MEDI528 30 mg vs MEDI528 100 mg vs MEDI528 300 mg; Combined MEDI-528 dose groups versus placebo; Test type: Superiority or Other; p = 0.574, Fisher Exact

17. Secondary Outcome: Proportion of Participants With Detectable Anti-drug Antibodies to MEDI-528
Description: Proportion of participants with detectable anti-drug antibodies to MEDI-528 in subjects receiving 30, 100, or 300 mg MEDI-528 and placebo
Time Frame: Days 1, 29, 57, 85, 127, 169, 176, 204,260, and 323
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81), or placebo (n=82) group and received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 82 | 81 | 83 | 81
Participants | 4 | 15 (1.53) | 4 (1.83) | 3 (1.99)

18. Secondary Outcome: First Dose Trough Concentration of MEDI-528
Description: First dose trough concentration of MEDI-528 measured on Day 15 prior to administration of the second dose of MEDI-528 (30, 100, or 300 mg). Serum concentrations of MEDI-528 were measured on Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323. The first dose trough concentration of MEDI-528 was measured on Day 15 prior to the Day 15 dose.
Time Frame: Day 15
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 group (n=81, 83, or 81, respectively).
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 0 | 81 | 83 | 81
Microgram per milliliter |  | 2.15 (0.81) | 5.91 (2.97) | 15.80 (5.68)

19. Secondary Outcome: Day 169 Steady State Trough Concentration of MEDI-528
Description: Trough concentration of MEDI-528 measured on Day 169 prior to administration of the last dose of MEDI-528 (30, 100, or 300 mg). Serum concentrations of MEDI-528 were measured on Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323. Steady state trough concentration of MEDI-528 was measured on Day 169.
Time Frame: Day 169
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 group (n=81, 83, or 81, respectively).
Measure: Mean (Standard Deviation); unit: Microgram per milliliter
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 0 | 81 | 83 | 81
Microgram per milliliter |  | 5.99 (3.37) | 21.68 (9.49) | 61.57 (26.85)

20. Secondary Outcome: Half Life of MEDI-528
Description: Half life of MEDI-528 in subjects receiving 30, 100, or 300 mg MEDI-528. Serum concentrations of MEDI-528 were measured on Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323.
Time Frame: Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323
Population: All participants randomized into the 30, 100, or 300 mg MEDI-528 group (n=81, 83, or 81, respectively).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 0 | 81 | 83 | 81
Days |  | 39.0 (8.14) | 32.6 (5.89) | 32.2 (6.41)

21. Secondary Outcome: Accumulation Ratio of Trough Concentrations of MEDI-528
Description: Accumulation ratio of trough concentrations of MEDI-528 in subjects receiving 30, 100, or 300 mg MEDI-528. Serum concentrations of MEDI-528 were measured on Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323.
Time Frame: Days 1, 15, 29, 57, 85, 127, 169, 176, 204, 232, 260, 288, and 323
Population: All participants who were randomized into the 30 mg MEDI-528 (n=81), 100 mg MEDI-528 (n=83), 300 mg MEDI-528 (n=81) and received at least one dose of investigational product.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Number analyzed (Participants) | 0 | 81 | 83 | 81
Ratio |  | 3.46 (1.53) | 4.18 (1.83) | 4.11 (1.99)

ADVERSE EVENTS:
Time Frame: Day 1 to Day 323
Arm/Group | Placebo | MEDI528 30 mg | MEDI528 100 mg | MEDI528 300 mg
Serious Adverse Events (participants affected / at risk) | 4/82 | 9/81 | 4/83 | 2/81
Other Adverse Events (participants affected / at risk) | 67/82 | 62/81 | 68/83 | 69/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | MEDI528 30 mg (N=81) | MEDI528 100 mg (N=83) | MEDI528 300 mg (N=81)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lobar pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Complicated migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=82) | MEDI528 30 mg (N=81) | MEDI528 100 mg (N=83) | MEDI528 300 mg (N=81)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (4) | 3 (3)
Toothache (Gastrointestinal disorders) | 1 (1) | 2 (2) | 4 (4) | 0 (0)
Asthenia (General disorders) | 2 (3) | 3 (3) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 2 (3) | 1 (2) | 4 (10) | 5 (9)
Injection site pain (General disorders) | 5 (6) | 1 (1) | 4 (5) | 2 (14)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Acute sinusitis (Infections and infestations) | 2 (2) | 3 (4) | 2 (2) | 2 (4)
Bronchitis (Infections and infestations) | 8 (8) | 4 (5) | 2 (3) | 5 (7)
Gastroenteritis (Infections and infestations) | 3 (3) | 2 (2) | 5 (5) | 2 (2)
Influenza (Infections and infestations) | 6 (8) | 10 (11) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 12 (15) | 11 (15) | 5 (9) | 7 (11)
Pharyngitis (Infections and infestations) | 2 (2) | 4 (4) | 8 (13) | 4 (5)
Rhinitis (Infections and infestations) | 5 (5) | 3 (3) | 3 (3) | 2 (2)
Sinusitis (Infections and infestations) | 4 (5) | 10 (11) | 4 (4) | 6 (10)
Upper respiratory tract infection (Infections and infestations) | 12 (19) | 6 (6) | 16 (23) | 20 (32)
Urinary tract infection (Infections and infestations) | 6 (6) | 7 (9) | 7 (7) | 2 (3)
Viral upper respiratory tract infection (Infections and infestations) | 5 (7) | 1 (4) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 3 (3) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 3 (4)
Dizziness (Nervous system disorders) | 5 (5) | 2 (2) | 5 (15) | 0 (0)
Headache (Nervous system disorders) | 8 (11) | 13 (20) | 5 (9) | 6 (7)
Migraine (Nervous system disorders) | 1 (1) | 4 (5) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 25 (41) | 28 (53) | 20 (29) | 31 (64)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 1 (1) | 3 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 2 (2) | 1 (2) | 4 (5)
Hypertension (Vascular disorders) | 2 (3) | 4 (4) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.